CLINICAL TRIAL: NCT06759727
Title: Outcomes of Different Surgical Procedures After High Level Resection for Patients With Small Intestinal Gangrene
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Shendy Abdelsayed, resident, Assiut University
Other Study IDs: small bowel gangrene surgery
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Small Bowel Gangrene; Mesenteric Artery Ischemia; Strangulated Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — parts of small intestine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: Primary anastomosis: using hand sewing technique
- Group B: Primary anastomosis with prophylactic tube enterostomy. Feeding jejunostomy may be inserted
- Group C: Jejunostomy: double barrel stoma.
- Group D: Jejunostomy: double barrel stoma with distal refeeding via the mucous fistula opening.

SUMMARY:
In this cohort study, aim to evaluate and compare short-term postoperative outcomes of different surgical procedures for patients with intestinal gangrene who underwent high level small bowel resection (< 150 cm from DJ).

DETAILED DESCRIPTION:
Patients with intestinal gangrene have a high mortality rate depending on etiology, degree, and length of an ischemic part, associated comorbidity, and time between the onset of symptoms and final diagnosis. This overall mortality ranges from 50 to 80%. When intestinal gangrene is evident or suspected, surgical laparotomy is mandatory, where the affected segment is resected, and the remaining part is either anastomosed or diverted on the anterior abdominal wall as stoma.

Small bowel anastomoses performed in the emergency settings have a high risk of anastomotic leakage. The leak rate in these settings may reach 35% . Intestinal gangrene is usually associated with peritonitis and sepsis. The performance of ostomy or intestinal anastomosis in cases of peritonitis or sepsis is a controversial theme. This controversy increases when proximal small bowel is involved .

Stomas avoid the risks of anastomotic leakage and re-operation and permit close examination of the bowel by inspection. However, creating stoma after proximal level of resection is associated with catastrophic sequels of high output fistula and short bowel syndrome. Hence, most of the time the risk of a high jejunal anastomosis dehiscence is preferred to the metabolic complications associated with ostomy .

A jejunostomy was defined as having less than 200 cm of proximal remaining small bowel. Since most nutrients are absorbed within the first 100-150 cm of the jejunum, the severity of short bowel syndrome and dependence on TPN is markedly increased if a jejunostomy is created at less than 150 cm from DJ . Distal refeeding of chyme "re-feeding enteroclysis", by reinfusing the chyme collected from the proximal stoma into the downstream small bowel through the distal stoma, was used by some surgeons to alleviate the complications of jejunostomy before re-establishment of digestive continuity . However, this procedure can be technically demanding. On the other hand, some authors prefer to use prophylactic tube enterostomy with primary anastomosis in cases of high risk of anastomotic leak .

The choice between these surgical technical varieties depends upon general health status of the patient, and local abdominal factors e.g. presence of peritoneal contamination, but mostly depends on surgeons' experience.

ELIGIBILITY:
Inclusion Criteria:

* 1) Distance of proximal resection margin less than 150 cm from DJ. 2) Mesenteric vascular ischemia. 3) Strangulating obstruction e.g. due to hernia, volvulus, band, etc.

Exclusion Criteria:

* 1) Patients less than 18 years. 2) Patients with malignant disease. 3) Patients with almost all small bowel loops resected (< 60 cm remaining).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective non-randomized comparative study. Patients who will undergo high level small bowel resection for intestinal gangrene during the period from September 2024 to September 2026 are included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
morality rate | within 90 days of surgery